CLINICAL TRIAL: NCT04936490
Title: Efficacy and Safety of Crocin Supplementation in Patients With Central Serous Chorioretinopathy (CSCR)
Brief Title: Crocin Supplementation in CSCR
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mojtaba Heydari, Principal Investigator, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1400.059
Record Dates: First submitted 2021-05-02; First posted 2021-06-23 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Chorioretinopathy, Central Serous
MeSH Terms: conditions — Central Serous Chorioretinopathy | interventions — crocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crocin (Experimental)
  Interventions: Drug: Crocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Crocin — 15 mg/d
  Arms: Crocin
Drug: Placebo — 15 mg/d
  Arms: Placebo

SUMMARY:
Preclinical and clinical evidence support the protective effect of crocin on different pathologic pathways involved in central serous chorioretinopathy (CSCR). They involve inflammation, oxidative stress, mineralocorticoid pathway, and also stress-related injuries. It also showed that crocin has a protective effect on the retinal pigmented epithelium (RPE) layer. Based on the mentioned evidence the study designed to evaluate the efficacy and safety of 2-month crocin supplementation (15 mg/d) in 40 patients with CSCR in a randomized controlled blinded clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-60 years old
* The diagnosis of CSCR based on clinical and imagining evaluation
* informed consent

Exclusion Criteria:

* Chronic CSCR
* Laser treatment (6 months prior to enrollment)
* IVB treatment (3 months prior to enrollment)
* Other retinal diseases
* History of eye diseases
* Diabetes Mellitus
* Renal or hepatic diseases
* Allergy to saffron or crocin
* Pregnancy or lactation
* Beta-blocker, diuretic, or corticosteroid (1 week prior to enrollment) Bleeding tendency or any coagulation disorder

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Best-corrected visual acuity (BCVA) | 8 weeks

SECONDARY OUTCOMES:
Foveal thickness (μm) | 8 weeks
  measured by OCT imaging
Subretinal fluid height (μm) | 8 weeks
  measured by OCT imaging
Subfoveal choroidal thickness (μm) | 8 weeks
  measured by OCT imaging
Number of participants need to laser therapy | 8 weeks
  based on clinical criteria
Total number of reported adverse events | 8 weeks
  based on patients reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran